CLINICAL TRIAL: NCT00025324
Title: Clinical Correlative Studies In Primary Central Nervous System Germ Cell Tumors: The Third International CNS Germ Cell Tumor Study Group Protocol
Brief Title: Chemotherapy, Surgery, Radiation Therapy and Bone Marrow or Peripheral Stem Cell Transplantation in Treating Patients With Primary CNS Germ Cell Tumors
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Children's Hospital Los Angeles (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000068950; CHLA-NYU-0007H; NCI-G01-2019
Record Dates: First submitted 2001-10-11; First posted 2003-01-27 (Estimated); Last update posted 2013-12-18 (Estimated); Status verified 2004-12

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: childhood central nervous system germ cell tumor; adult central nervous system germ cell tumor
MeSH Terms: conditions — Central Nervous System Neoplasms | interventions — Filgrastim; Carboplatin; Cyclophosphamide; Etoposide; Thiotepa; Peripheral Blood Stem Cell Transplantation; Radiotherapy

INTERVENTIONS:
Biological: filgrastim
Drug: carboplatin
Drug: cyclophosphamide
Drug: etoposide
Drug: thiotepa
Procedure: autologous bone marrow transplantation
Procedure: bone marrow ablation with stem cell support
Procedure: conventional surgery
Procedure: peripheral blood stem cell transplantation
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Peripheral stem cell transplantation or bone marrow transplantation may allow the doctor to give higher doses of chemotherapy drugs and kill more tumor cells. Radiation therapy uses high-energy x-rays to damage tumor cells.

PURPOSE: Phase II trial to study the effectiveness of chemotherapy, surgery, radiation therapy, and bone marrow or peripheral stem cell transplantation in treating patients who have primary CNS germ cell tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the two-year event-free survival of patients with primary CNS germ cell tumors treated with carboplatin, etoposide, cyclophosphamide, and filgrastim (G-CSF) with or without radiotherapy and/or high-dose chemotherapy with autologous bone marrow or peripheral blood stem cell transplantation.
* Determine the prognostic significance of slow-responding tumor marker normalization in patients treated with this regimen.
* Determine the prognostic significance of syncytiotrophoblastic giant cell component and cerebrospinal fluid beta-human chorionic gonadotropin elevation in patients treated with this regimen.
* Assess the early and late endocrinologic, neuropsychometric, and quality of life sequelae in patients treated with this regimen.

OUTLINE: This is a multicenter study. Patients are stratified according to risk status (low vs intermediate or high).

Regimen A (Low-risk patients)

* Chemotherapy: Patients receive carboplatin IV over 4 hours and etoposide IV over 2 hours on days 1-2 and filgrastim (G-CSF) subcutaneously (SC) once daily beginning on day 3 and continuing until blood counts recover (course 1). Patients also receive cyclophosphamide IV over 1 hour and etoposide IV over 2 hours on days 22 and 23 and G-CSF SC once daily beginning on day 24 and continuing until blood counts recover (course 2).
* Patients with complete response (CR) to initial chemotherapy receive 2 additional courses of chemotherapy as above and then proceed to observational phase. Patients with partial response (PR) to initial chemotherapy receive 2 additional courses of chemotherapy as above.
* Patients with CR after additional chemotherapy receive another 2 additional courses of chemotherapy as above and then proceed to observational phase. Patients with PR after additional chemotherapy undergo biopsy and/or resection of residual tumor.
* Patients with evidence of malignant germ cell tumor (GCT) on resection undergo radiotherapy. Patients with no evidence of malignant GCT on resection but with scar, fibrosis, or mature teratoma receive 2 additional courses of chemotherapy as above and then proceed to observational phase. Patients with no evidence of malignant GCT on resection but with immature teratoma receive carboplatin IV over 4 hours, cyclophosphamide IV over 1 hour, and etoposide IV over 2 hours on days 1-2 and 22-23. Patients who underwent complete resection of residual tumor proceed to observational phase. Patients who underwent a biopsy only or an incomplete resection of residual tumor undergo radiotherapy.

Regimen B (Intermediate and high-risk patients)

* Patients receive carboplatin IV over 4 hours, cyclophosphamide IV over 1 hour, and etoposide IV over 2 hours on days 0-1. Patients also receive G-CSF SC once daily beginning on day 2 and continuing until blood counts recover. Treatment repeats every 21 days for a total of 2 courses. Patients undergo bone marrow or peripheral blood stem cell harvest prior to second course of chemotherapy.
* Patients with rapid CR to 2 initial courses of chemotherapy receive an additional 2 courses of chemotherapy as above and then proceed to observational phase. Patients with a PR or slow response to 2 initial courses of chemotherapy receive 2 additional courses of chemotherapy as above. Patients with a CR to courses 3 and 4 receive 2 more courses of chemotherapy and then proceed to observational phase. Patients with a PR to courses 3 and 4 undergo a biopsy and/or resection of residual tumor.
* Patients with no evidence of malignant GCT on resection but with scar, fibrosis, or mature teratoma receive carboplatin IV over 4 hours and etoposide IV over 2 hours on days 1 and 2 and cyclophosphamide IV over 1 hour and etoposide IV over 2 hours on days 22 and 23 and proceed to observational phase. Patients with teratoma on resection receive additional treatment as in regimen A. Patients with evidence of pure germinoma on resection undergo radiotherapy.
* Patients with evidence of other malignant GCT on resection undergo high-dose chemotherapy (HDCx) with bone marrow or peripheral blood stem cell support (PBSCS) comprising thiotepa IV over 3 hours and etoposide IV over 1 hour on days -8 through -6; carboplatin IV over 4 hours on days -5 through -3; reinfusion of autologous bone marrow or peripheral blood stem cells on day 0; and G-CSF SC or IV every 12 hours beginning on day 1 and continuing until blood counts recover. Patients then undergo radiotherapy.

Quality of life is assessed before bone marrow or PBSCS and then every 2 years thereafter.

Patients are followed at day 42, at 3 months, then every 3 months for 1 year, every 4 months for 1 year, every 6 months for 3 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 80 patients (40 per stratum) will be accrued for this study within 4 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed newly diagnosed primary CNS germ cell tumor OR
* Serum or cerebrospinal fluid (CSF) elevation of alpha-fetoprotein (AFP) or beta-human chorionic gonadotropin (beta-HCG) greater than 50 ng/mL
* Low-risk disease:

  * Histologically proven pure germinoma
  * Localized, nonmetastatic disease
  * Normal CSF
  * Normal serum tumor markers
* Intermediate-risk disease:

  * Histologically proven germinoma
  * Beta-HCG-positive syncytiotrophoblastic giant cell component AND/OR
  * CSF elevation of beta-HCG to less than 50 ng/mL
* High-risk disease:

  * Histologically proven choriocarcinoma, endodermal sinus tumor, or embryonal carcinoma
  * Elevated serum and/or CSF AFP OR
  * Elevated serum beta-HCG OR
  * Elevated CSF beta-HCG greater than 50 ng/mL OR
  * Disseminated disease by MRI and/or CSF cytology

PATIENT CHARACTERISTICS:

Age:

* Any age

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Bilirubin less than 2.0 mg/dL
* Indirect hyperbilirubinemia due to Gilbert's syndrome is allowed
* AST and ALT less than 5 times upper limit of normal

Renal:

* Creatinine clearance greater than 60 mL/min

Cardiovascular:

* Cardiac function normal by echocardiogram
* No myocardial infarction or ischemia in patients over 30 years
* Fractional shortening greater than 30%

Other:

* No unacceptable morbidity of organ systems outside the CNS
* Not pregnant
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No prior chemotherapy

Endocrine therapy:

* No concurrent corticosteroids administered solely for antiemesis during study chemotherapy

Radiotherapy:

* No prior cranial radiotherapy

Surgery:

* Not specified

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2000-12

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan L. Finlay, MB, ChB, Study Chair — Children's Hospital Los Angeles
Locations (4):
- United States (2):
  - Children's Hospital Los Angeles, Los Angeles, California
  - Children's Hospital of the King's Daughters, Norfolk, Virginia
- Princess Margaret Hospital for Children, Perth, Western Australia, Australia
- Tom Baker Cancer Centre - Calgary, Calgary, Alberta, Canada